CLINICAL TRIAL: NCT02748031
Title: Congenital Cataract Morphological Classifications and Monitoring Using Slit-Lamp-Adapted Photography in CCPMOH
Brief Title: Congenital Cataract Morphological Classifications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Erping Long, Principal Investigator，Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCPMOH2016-China4
Record Dates: First submitted 2016-04-17; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Congenital Cataract
Keywords: Congenital cataracts; Opacity location; Opacity shape; Classification; Clinical applicability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eligible patients group (Experimental)
  Interventions: Procedure: slit-lamp-adapted anterior segmental photography

INTERVENTIONS:
Procedure: slit-lamp-adapted anterior segmental photography — The eligible patients underwent pupil dilation and slit-lamp-adapted anterior segmental photography to electronically record and monitor the morphology of their cataractous lens.

SUMMARY:
Photography is considered as one of the most important means to promote evidence-based medical practice in pediatric ophthalmology.This study is to investigate the feasibility of congenital cataract morphological classifications and monitoring using slit-lamp-adapted anterior segmental photography in a large cohort that included uncooperative children.

DETAILED DESCRIPTION:
Lens opacities in congenital cataracts have a wide range of presentations.Therefore, it is important to find a method of recording, classifying and monitoring cataract morphologies that is feasible and safe in a large cohort of children with congenital cataracts, including uncooperative children. Photography is considered as one of the most important means to promote evidence-based medical practice in pediatric ophthalmology.

In this study, the investigators studied congenital cataract morphological classifications and monitoring using slit-lamp-adapted anterior segmental photography and evaluated its safety and feasibility in pediatric cataract patients registered in the Childhood Cataract Program of the Chinese Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* Children with pediatric unilateral/bilateral cataracts
* Children who were younger than 10 years of age

Exclusion Criteria:

* Premature birth
* Microphthalmia
* Micro-or Megalocornea
* Keratoconus
* Glaucoma
* Traumatic or complicated cataracts
* Vitreous and retinal diseases
* Any previous surgeries, and contraindication for pupil dilation and sedation

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1050 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Congenital Cataract Morphological Classifications and Monitoring using Slit-Lamp-Adapted Photography | baseline
  All eligible pediatric patients underwent pupil dilation with compound tropicamide eye drops 3 times (1 time every 10 minutes) before the examination or administration of sleep aid medicine. Then, the children underwent slit-lamp-adapted anterior segmental photography (BX900, Haag-Streit AG, Köniz, Switzerland) for each cataractous lens, including one diffuse light photo, one slit-light photo across the cataract and one retro-illumination photo. All photos of the included patients were screened and morphologically classified separately by two pediatric ophthalmologists; a third ophthalmologist was masked and required to make a decision if the first two physicians had different opinions.

CONTACTS AND LOCATIONS:
Overall Officials: Hantian Lin, M.D., Ph.D, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Erping Long, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lin H, Chen W, Luo L, Congdon N, Zhang X, Zhong X, Liu Z, Chen W, Wu C, Zheng D, Deng D, Ye S, Lin Z, Zou X, Liu Y. Effectiveness of a short message reminder in increasing compliance with pediatric cataract treatment: a randomized trial. Ophthalmology. 2012 Dec;119(12):2463-70. doi: 10.1016/j.ophtha.2012.06.046. Epub 2012 Aug 24. PMID 22921386
- [Derived] Long E, Lin Z, Chen J, Liu Z, Cao Q, Lin H, Chen W, Liu Y. Monitoring and Morphologic Classification of Pediatric Cataract Using Slit-Lamp-Adapted Photography. Transl Vis Sci Technol. 2017 Nov 2;6(6):2. doi: 10.1167/tvst.6.6.2. eCollection 2017 Nov. PMID 29134133
- See also: Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/